CLINICAL TRIAL: NCT00661583
Title: Occlusion Prevention for Trabeculectomy Procedures Using Combination Ranibizumab and Mitomycin C (MMC) During Surgery (OCTOPUS Study)
Brief Title: Use of Ranibizumab With Mitomycin C During Trabeculectomy
Acronym: OCTOPUS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0921
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-08

CONDITIONS: Glaucoma
Keywords: trabeculectomy; glaucoma; ranibizumab
MeSH Terms: conditions — Glaucoma | interventions — Ranibizumab; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ranibizumab alone (Experimental): Treatment with ranibizumab 0.5 mg intravitreally injected (n=10)
  Interventions: Drug: Ranibizumab
- Ranibizumab and MMC (Experimental): Combination ranibizumab 0.5mg intravitreally injected and MMC (0.4 mg/ml for 2 min) in eyes after trabeculectomy (n=10)
  Interventions: Drug: Ranibizumab and MMC
- MMC alone (Active Comparator): MMC therapy alone (n=10)
  Interventions: Drug: MMC

INTERVENTIONS:
Drug: Ranibizumab — 0.5mg of ranibizumab intravitreally injected after surgery and at 1 month if needed
  Arms: Ranibizumab alone
Drug: Ranibizumab and MMC — Combination ranibizumab 0.5mg intravitreally injected and MMC (0.4 mg/ml for 2 min) in eyes after trabeculectomy
  Other Names: Ranibizumab and Mitomycin C
  Arms: Ranibizumab and MMC
Drug: MMC — MMC (0.4 mg/ml for 2 min) in eyes after trabeculectomy.
  Other Names: Mitomycin C
  Arms: MMC alone

SUMMARY:
The purpose of the study is to study the safety of the combination of ranibizumab and MMC vs monotherapy MMC vs intravitreal ranibizumab injection in patients with glaucoma.

DETAILED DESCRIPTION:
A common problem after undergoing trabeculectomy surgery to create a bleb (blister or bubble) to reduce intraocular pressure, is scarring of the opening. This scarring prevents fluid drainage and interferes with the proper functioning of the bleb. MMC (Mitomycin C) is usually administered intraoperatively, to reduce scarring and increase filtration. However, the failure rate of trabeculectomy remains high. Anti-VEGF (Vascular endothelial growth factor) agents have been used successfully in cases requiring bleb needling. The purpose of the study is to determine the safety of the combination of ranibizumab and MMC vs monotherapy MMC in patients with glaucoma.

This is an open-label, Phase I/II safety study of 30 patients randomized to either treatment with ranibizumab 0.5 mg intravitreally injected (n=10), combination ranibizumab 0.5mg intravitreally injected and MMC (0.4 mg/ml for 2 min) in eyes after trabeculectomy (n=10) or MMC therapy alone (n=10).

For the ranibizumab groups, a repeat injection of ranibizumab 0.5mg may be given PRN (as needed) at 1 month if hypervascularity or neovascularization of the conjunctiva exists.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma
* undergoing trabeculectomy
* 21 years of age or older

Exclusion Criteria:

* pregnancy or lactation
* any condition the investigator believes would impose a significant hazard to the patient if investigational therapy were initiated
* history of ocular surface disease
* cataract surgery in the past 6 months
* history of active inflammatory, infectious or idiopathic keratitis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malik Y. Kahook, MD, Study Director — Rocky Mountain Lions Eye institute
Locations (1):
- Rocky Mountain Lions Eye Institute, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Subject medical information obtained by this study is confidential, and disclosure to third parties other than those noted below is prohibited.
  Upon the subject's permission, medical information may be given to his/her personal physician or other appropriate medical personnel responsible for his/her welfare.
  Data generated by this study will be available for inspection upon request by representatives of the U.S. FDA, national and local health authorities, the drug manufacturer and the IRB/EC, if appropriate.

REFERENCES:
- [Derived] Kahook MY. Bleb morphology and vascularity after trabeculectomy with intravitreal ranibizumab: a pilot study. Am J Ophthalmol. 2010 Sep;150(3):399-403.e1. doi: 10.1016/j.ajo.2010.03.025. Epub 2010 Jun 8. PMID 20570237

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranibizumab Alone | Ranibizumab and MMC | MMC Alone
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab Alone | Ranibizumab and MMC | MMC Alone | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 2 | 11
  Male | 4 | 7 | 8 | 19
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Ocular Adverse Events
Description: To assess ocular adverse events of combination ranibizumab and MMC therapy at 6 months
Time Frame: 6 months
Measure: Number; unit: Number of Reported Adverse Events
Arm/Group | Ranibizumab Alone | Ranibizumab and MMC | MMC Alone
Number analyzed (Participants) | 10 | 10 | 10
Number of Reported Adverse Events | 0 | 0 | 0

2. Secondary Outcome: Percent of Subjects With a Qualified Success and Viable Bleb at 6 Months.
Description: To determine percent of subjects with a qualified success and viable bleb at 6 months (IOP between 6mm Hg and 22 mm Hg with pressure controlled with and without adjunctive medications)
Time Frame: 6 months
Measure: Number; unit: percentage of subjects
Arm/Group | Ranibizumab Alone | Ranibizumab and MMC | MMC Alone
Number analyzed (Participants) | 10 | 10 | 10
percentage of subjects | 100 | 100 | 100

3. Secondary Outcome: Mean Change in in Intraocular Pressure.
Description: Mean change in in intraocular pressure at 3 months and at 6 months
Time Frame: 6 months
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Ranibizumab Alone | Ranibizumab and MMC | MMC Alone
Number analyzed (Participants) | 10 | 10 | 10
mmHg
  month 3 minus baseline | -6.40 [-26 to 2] | -6.40 [-15 to 0] | -8.35 [-26 to 0]
  month 6 minus baseline | -6.60 [-32 to -1] | -4.90 [-16 to 1] | -8.00 [-24 to -2]

4. Secondary Outcome: Mean Change in Visual Acuity
Description: Mean change in visual acuity in logMAR.
Time Frame: 6 months
Measure: Mean (Full Range); unit: logMAR
Arm/Group | Ranibizumab Alone | Ranibizumab and MMC | MMC Alone
Number analyzed (Participants) | 10 | 10 | 10
logMAR
  Month 3 minus baseline | -0.01 [-0.22 to 0.12] | 0.01 [-0.12 to 0.18] | 0.13 [-0.04 to 0.48]
  Month 6 minus baseline | -0.05 [-0.22 to 0.13] | 0.05 [-0.14 to 0.18] | 0.13 [-0.05 to 0.32]

ADVERSE EVENTS:
Arm/Group | Ranibizumab Alone | Ranibizumab and MMC | MMC Alone
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No